# Universidad de California, San Diego Consentimiento para Participar como Sujeto en Investigación

"LinkUP": Es una intervención conductual dentro del Proyecto "Etno-epidemiologia de Hepatitis C, (VHC), VIH y sobredosis asociados con el Narcomenudeo y Turismo de Drogas", también conocido como Proyecto "La Frontera".

#### Introducción

La Dra Steffanie Strathdee, Ph.D.y la Coalición de Reducción del Daño de San Diego (HRCSD, "OnPoint") están realizando esta investigación y le están solicitando su consentimiento para participar. Este estudio ha recibido fondos de los Institutos Nacionales de Salud y de la Aceleración Rápida de Diagnostico en Poblaciones Carentes (RADxUP). Esta sección le brindara un resumen de la información más importante. El resto del documento le brindará mas detalles.

- La investigación es voluntaria ya sea si Ud. se suma o no es su decisión. Ud. puede comentar su decisión con otros (como sería su familia y amistades).
- Ud. puede estar de acuerdo ahora y cambiar de opinión después.
- Si Ud. se niega a participar, no lo tomaremos en su contra.
- Su decisión no afectara ninguno de los otros beneficios a los que ya tiene derecho.
- Por favor, haga todas las preguntas y manifieste sus preocupaciones antes, durante y después de la investigación.

**Resúmen**: Estamos realizando esta investigación para ver si el combinar educación, entrevista motivacional y resolución de problemas aumenta el hacerse la prueba de COVID-19 y la vacunación contra el COVID-19 en personas que se inyectan drogas y que asisten a los programas de intercambio de jeringas. Se le pedirá que participe en una sesión breve educacional y o conductual y luego se le ofrecerá hacerse la prueba de COVID-19 y se lo referirá a una clínica cercana que le pueda ofrecer la vacuna contra el COVID-19. También se le pedirá que complete una entrevista suplementaria.

**Beneficios**: Su participación en este estudio nos podría ayudar a aprender por qué algunas personas demoran el hacerse la prueba de COVID-19 o el vacunarse y sobre los efectos de COVID-19 en personas que se inyectan drogas. Nosotros esperamos poder usar esta información llevar a cabo investigación relacionada a la salud y conducta en personas que se inyectan drogas, lo que eventualmente se puede utilizar para diseñar intervenciones apropiadas y efectivas y programas de salud en su comunidad.

**Riesgos**: Los riesgos más comunes esperados en el estudio tienen que ver con el platicar sobre temas que lo puedan hacer sentir incomodo o molesto. Ud. le puede pedir a cualquiera de los investigadores o consejeros de OnPoint que se retiren, dejen de hablarle en cualquier momento y puede cambiar de opinión sobre su participación en el estudio

LinkUP aun cuando se haya empezado la sesión. Si Ud. desea ver a un consejero después de platicar con nosotros, podemos hacer los arreglos necesarios sin ningún costo para Ud.

El riesgo más serio del estudio incluye la perdida de confidencialidad. Aunque en ningún momento sus respuestas o resultados individuales que incluyan su nombre estarán disponibles a ninguna persona ajena al Proyecto, existe una mínima posibilidad que alguien pudiera descubrir que Ud. ha participado en el proyecto. Si esto llegara a ocurrir, podría afectar su empleo y/o seguranza. Los miembros de nuestro equipo harán todo el esfuerzo necesario para proteger su confidencialidad y le darán las referencias apropiadas a las autoridades de salud locales para su atención. También le brindaremos una tarjeta del estudio y un número gratuito 1-800 para que nuestro equipo de investigación pueda abogar en su representación en caso necesario.

A continuación, se ofrece más información adicional. Por favor con toda libertad haga las preguntas que desee antes de firmar el consentimiento.

# ¿Qué es INS y RADxUP?

INS quiere decir Institutos Nacionales de Salud. El INS forma parte del Departamento de Servicios Humanos y de Salud de los Estados Unidos. El propósito de INS es el de descubrir nuevos conocimientos que puedan llevar a una mejor salud para todos. El INS ha otorgado los fondos (brindado recurso) para el programa RADxUP. En la parte de San Diego a este programa lo llamamos estudio LinkUP.

RADx-UP quiere decir Aceleración Rápida de Diagnostico en Poblaciones Carentes. RADx-UP programa de investigación en salud para aprender más sobre el COVID-19. Si Ud. se une al Proyecto Link-UP, nosotros recolectaremos datos (información) sobre Ud. Nosotros combinaremos estos datos con los de otras personas que se unirán a RADx-UP sin su nombre o sin cualquier otra información adjunta que permita identificación personal. Nosotros estudiaremos los datos de todas las personas que se unan a al estudio para entender cómo se podría ayudar más a las personas en riesgo de contraer o que ya tengan COVID-19.

# ¿Por qué se le está pidiendo que participe, cómo se lo seleccionó y cuál es la cantidad aproximada de participantes en el estudio?

Se le está pidiendo que participe en LinkUP porque Ud. ya está reclutado en el Proyecto La Frontera, y Ud.: a) tiene al menos 18 años de edad; b) es residente del condado de San Diego County donde se está realizando este estudio; c) Ud. indicó en su entrevista de seguimiento que nunca se hizo la prueba de COVID-19 de manera voluntaria fuera de La Frontera; d) y que Ud. se ha vacunado con dos o menos dosis contra el COVID-19, siendo la aplicación de la última dosis hace más de 6 meses; e) estuvo de acuerdo en compartir su expediente médico con el equipo del estudio LinkUP; y f) estuvo de acuerdo en ser contactado para este estudio. Se invitará a participar en LinkUP a otras 149 personas más.

# ¿Qué le pasará en el estudio y cuáles procedimientos son estándar de atención y cuáles son experimentales?

Si Ud. decide unirse al estudio LinkUP y si Ud. ha completado su última visita de seguimiento de La Frontera hace más de 3 meses, el personal de La Frontera le pedirá que complete una entrevista con preguntas sobre su estilo de vida, actitudes, comportamientos, problemas de salud y si se ha hecho la prueba de COVID-19 y si se ha vacunado contra el COVID-19. Se le compensará con \$20 dólares por esta visita.

A continuación, el personal de La Frontera le entregará un cupón enmicado con la dirección y horarios de los sitios más cercanos donde se encuentra el programa de Intercambio de Jeringas OnPoint. El asistir a los sitios de OnPoint es voluntario. OnPoint programa de intercambio de jeringas que ofrece servicios gratuitos en varios lugares en los alrededores del condado de San Diego, y que incluye la prueba de COVID-19 y referencias para sitios de vacunación contra el COVID-19 como estándar de atención. Cuatro de estos lugares de atención participaran en el estudio LinkUP. En dos de los 4 lugares, se les ofrecerá a los participantes de LinkUP educación sobre COVID-19 solamente y en los otros dos lugares, se les ofrecerá a los participantes de LinkUP consejería con entrevista motivacional (EM) sobre COVID-19.

Si Ud. visita el lugar de OnPoint, sus consejeros le asignarán un identificador único (IU) si Ud. nunca antes había usado sus servicios. Estos IU se generan usando las 1&3 letras de primer nombre y del apellido, fecha de nacimiento, e identificador de sexo equivalente a H-1, M-2, Otro-3.

Los consejeros pares de OnPoint le harán una breve entrevista de 5 minutos sobre COVID-19, que incluirá información sobre cualquier síntoma (cambio en u estado de salud) y resultados de sus pruebas. Si Ud. tuvo una prueba positiva al COVID-19, le pedirán información sobre rastreo de contactos (personas con las que Ud. pueda haber estado en contacto mientras Ud. tenía COVID-19). Le preguntarán sobre su historia médica y si Ud. se ha vacunado o no y por qué.

Luego, el consejero par de OnPoint le platicará sobre COVID-19, e incluirá información sobre el virus, como se transmite, que tipo de problemas de salud provoca y cuales vacunas y tratamientos hay disponibles para el virus. Ellos también le comentaran si alguna de la información que Ud. escucho sobre el COVID-19 o sobre las vacunas contra el COVID es correcta y cual información es incorrecta. Dependiendo del lugar de OnPoint que Ud. este visitando, el consejero podría platicar con Ud. sobre sus preocupaciones sobre COVID-19 y las vacunas. Los consejeros de OnPoint responderán cualquier pregunta que Ud. tenga. Sin importar que lugar de OnPoint Ud. visite, esta sesión se completara dentro de 45 minutos.

El consejero le ofrecerá a Ud. las pruebas de COVID-19 como estándar de atención. Ud. se puede rehusar a participar en la intervención LinkUP y aun así tener acceso a la prueba rápida para COVID-19 de antígenos gratuita (BiNaxNow®) en los programas de

Sitio del Estudio: San Diego

intercambio de jeringas en todo California, incluyendo OnPoint. Esto es distribuido por el Departamento de Salud Pública de California (CPHD). Para la vacunación gratuita contra el COVID-19 se le dará una referencia para las clínicas cercanas.

Si Ud. decide hacerse la prueba rápida de antígenos de COVID-19, el consejero le entregara sus resultados en 15 minutes. Si su prueba es positive, se le pedirá que se haga un hisopado nasal para una prueba confirmatoria de PCR. Ud. se puede rehusar a realizarse esta otra prueba si lo desea. La prueba de PCR de su hisopado nasal se realizará en un laboratorio certificado dentro de los próximos siguientes días. Si Ud. le da su información de contacto al consejero, ellos se pondrán en contacto con Ud. para compartirle los resultados de la prueba. Si Ud. sale positive para COVID-19 en cualquiera de estas pruebas o si tiene síntoma, será referido a su proveedor de salud para su seguimiento y se debería aislar de los demás. Si Ud. siente que no tiene un lugar seguro donde asilarse, el consejero lo podría referir a un albergue. Si su prueba es negativa para el virus que causa el COVID-19, el virus no se ha detectado. Sin embargo, es posible que Ud. reciba un resultado falso negativo por lo que Ud. podría tener COVID-19. Si Ud. está preocupado que pueda tener COVID-19, el consejero lo referirá a un proveedor de salud.

Si Ud. decide ponerse una de las vacunas contra el COVID-19 aprobadas por la ADA como seria Pfizer, Moderna y Janssen, Ud. poner obtener mas información por parte del personal en los programas de intercambio de jeringas de OnPoint como estándar de atención. La vacuna se pone con una jeringa en el brazo.

### ¿Cuánto tiempo durará cada procedimiento del estudio?

Si Ud. ha completado su última visita de seguimiento de La Frontera hace más de 3 meses y ahora debe completar la entrevista conductual este proceso llevará unos 60 minutos. La entrevista de ingreso de OnPoint dura unos 10 minutos. La sesión de consejería de LinkUP durará unos 45 minutos.

Si Ud. decide hacerse la prueba de COVID-19 como estándar de atención, la prueba rápida demora unos 15 minutos y Ud. recibirá sus resultados ahí mismo. Si Ud. decide hacerse la prueba de COVID-19 de PCR, el hisopado nasal para la prueba dura unos 3 minutos, pero Ud. no recibirá los resultados hasta unos días después. Si Ud. le comparte su información de contacto al consejero, ellos se pondrán en contacto con Ud. para entregarle los resultados de su prueba de PCR.

# ¿Qué harán con mis datos?

Nosotros recolectaremos datos (información) sobre su sesión de consejería, si se hizo la prueba de COVID-19 en alguno de los lugares del programa de intercambio de jeringas de OnPoint si Ud. recibió la vacuna contra el COVID-19 después de visitar OnPoint. Nosotros obtendremos una parte de estos datos directamente de Ud. y que compartirá con

el personal de La Frontera. Para proteger su confidencialidad, realizaremos una vinculación de records sin utilizar información con nombres (es decir, basada solamente en su fecha de nacimiento y sexo, y esta combinación es exclusivamente suya).

Nosotros también recolectaremos información de otros lugares en donde Ud quizás recibió la prueba de COVID-19, vacuna o tratamiento. Ejemplos de este tipo de información que podríamos recolectar de otros lugares incluye, pero no se limita a ONPoint/Coalición de Reducción del Daño de San Diego, la base de datos de COVID-19 del Departamento de Servicios Humanos y de Salud de San Diego, acceso de expedientes de salud electrónicos de hospitales, programas de rehabilitación de drogas y del Centro para Servicios de MediCaid y Medicare, entre otros.

Aunque los datos no estarán vinculados con su nombre, nosotros mantendremos sus datos resguardados de manera segura (es decir con protecciones adicionales), junto con los datos de muchas otras personas que participaran en los programas RADxUP en todo el país. Los investigadores utilizaran estos datos para aprender más sobre el COVID-19 u otras enfermedades o condiciones.

El Instituto de Investigación Clínica de Duke (DCRI) es un grupo de investigación elegido por los Institutos Nacionales de Salud (INS) para combinar los datos recolectados por todos aquellos que participan en los estudios RADxUP.

El DCRI creara uno base de datos RADx-UP (sistemas que almacenan información electrónica).

Solo almacenara información no identificable que Ud. está de acuerdo en compartirnos.

- Se le asignara un código del estudio y a Ud. solo se lo identificara en la base de datos con ese código único.
- No incluirá su nombre ni ninguna otra información que lo pueda identificar a Ud. fácilmente.
- Nosotros planeamos transferir y mantener esos datos no identificables en una base de datos segura para investigación sobre COVID-19 en los INS. Otros investigadores podrían utilizar estos datos para estudios, aparte de los ya indicados en este consentimiento.
- Los investigadores solo tendrán acceso a sus datos no identificables y no podrán vincular los datos con Ud.
- Ya que los datos no se podrán vincular con Ud., nosotros no lo contactaremos para informarle o pedirle permiso dantes de compartir esos datos con los investigadores.

| Estoy de acuerdo en permitir a OnPoint y La Frontera que vinculen mis datos |
|-----------------------------------------------------------------------------|
| identificables v no identificables sin utilizar mi nombre. |

| Si | No |
|-----------|-------------------|
| Iniciales | <u>Inicial</u> es |

## ¿Qué riesgos están asociados con este estudio?

Existe la posibilidad de que se pierda la confidencialidad. Aunque en ningún momento los resultados individuales o las respuestas a las preguntas estarán disponibles para personas ajenas al estudio y los formularios del estudio no incluirán su nombre, existe una pequeña posibilidad de que alguien descubra que usted participó en este estudio. La información que permite identificarlo personalmente tales como su nombre y su dirección incluidas en la forma localizadora se mantendrán resguardados bajo llave en un archivero separado en las oficinas del proyecto solamente a disposición del personal del estudio. Es su elección si le dice o no a la gente que ha participado en este estudio. También existe una pequeña posibilidad que alguien se entere de las respuestas que dio en la intervención de LinkUP. Si esto sucediera, podría afectar sus posibilidades de empleo y/o seguridad.

Ya que este es un estudio de investigación, pueden existir otros riesgos desconocidos que no se pueden anticipar ahora. Los miembros de nuestro equipo estarán atentos y atenderán cualquier riesgo inesperado de manera oportuna. Se le informara a Ud. de cualquier hallazgo significativo que surja.

## ¿Cuáles son las alternativas para participar en este estudio?

Las alternativas para este estudio son no participar. Es su decisión el formar parte del estudio o no. Puede abandonar este estudio en cualquier momento. Si no desea responder una pregunta específica, no es necesario que lo haga. Si se retira del estudio, las Dras Harvey-Vera o Strathdee le preguntarán si desea retirar su consentimiento para utilizar la información recopilada hasta ese momento. Puede inspeccionar y hacer una copia de los registros de su participación en este proyecto. Ud. se puede rehusar a participar en la intervención LinkUP y aun así tener acceso a la prueba rápida para COVID-19 de antígenos gratuita (BiNaxNow®) en los programas de intercambio de jeringas en todo California, incluyendo OnPoint. Esto es distribuido por el Departamento de Salud Pública de California (CPHD).

## ¿Qué sucede si cambia de opinión acerca de participar?

Ud. puede abandonar este estudio en cualquier momento. Si no desea responder una pregunta específica, no es necesario que lo haga. Si se retira del estudio, las Dras Harvey-Vera o Strathdee le preguntarán si desea retirar su consentimiento para utilizar la información recopilada hasta ese momento. Puede inspeccionar y hacer una copia de los registros de su participación en este proyecto. Se le informara si se descubre cualquier información novel que pueda afectar su deseo de continuar en el estudio

¿Puede ser retirado del estudio sin su consentimiento?

Debido a la naturaleza de la investigación científica, el investigador puede retirarlo del estudio en cualquier momento. También puede ser retirado del estudio si no sigue las instrucciones que le dio el personal del estudio.

## ¿Se le compensará por participar en este estudio?

Si se le pide que complete la entrevista de comportamientos se le compensara con \$20 dólares al finalizar su entrevista de LinkUP. También se le compensará \$10 dólares cuando visite el sitio de OnPoint.

¿Existe algún costo asociado con la participación en este estudio? No habrá ningún costo para usted por participar en este estudio.

# ¿Qué pasa si se lesiona como resultado directo de participar en este estudio?

Si se lesiona como resultado directo de su participación en esta investigación, la Universidad de California le brindará la atención médica que necesite para tratar esas lesiones. La Universidad no le proporcionará ninguna otra forma de compensación si resulta lesionado. Puede llamar a la Oficina del Programa de Protección de Investigaciones Humanas al 858-246-HRPP (858-246-4777) para obtener más información sobre esto, para preguntar sobre sus derechos como sujeto de investigación o para informar problemas relacionados con la investigación.

## ¿Cómo protegerán mi privacidad?

Su privacidad es muy importante para nosotros. Nosotros tendremos mucho cuidado en proteger su privacidad. Sin embargo, siempre existe la posibilidad que, aun con los mayores esfuerzos, su identidad y/o su información recolectada durante el estudio puede ser liberada por accidente o ser vista por personas no autorizadas. A continuación, describimos las medidas que tomaremos:

- Todos los que trabajan en este estudio han sido capacitados para respetar la privacidad de los participantes del estudio. Nunca discutirán lo que les ha dicho de una manera que pueda identificarlo.
- Su nombre u otra información de identificación no estará en ninguna nota o dato. Este formulario de consentimiento y la localizadora serán los únicos formularios con su nombre. Se guardarán en la Universidad de California, San Diego, EUA, en un cajón con llave. Nunca revelaremos que participó o cualquier otra información sobre su visita a nadie más, en la medida en que la ley nos lo permita. La información de su encuesta se etiquetará solo con un número de estudio y no con su nombre.
- Los datos se mantendrán almacenados en sistemas de computadoras encriptados, seguros y protegidos. Nosotros limitaremos y mantendremos una bitácora de quien puede acceder a estos datos. Nuestro equipo del estudio utilizara computadoras de nuestro departamento de sistemas de salud de UCSD, equipados con programas contra virus y malware, chips de seguridad TPM, y se conectaran por VPN.

- Cualquiera que pueda ver los datos necesitara tener una clave.
- Nosotros implementaremos estos pasos para proteger su información de otros que no deberían tener acceso a esos datos.
- Cuando sus datos sean compartidos con otros investigadores, no incluirán información que lo pueda identificar.
- Después de dicha eliminación, la información podría usarse para estudios de investigación futuros o distribuirse a otro investigador para estudios de investigación futuros sin su consentimiento informado adicional.

Esta investigación estará cubierta por un Certificado de Confidencialidad de los Institutos Nacionales de Salud. Los investigadores con este Certificado no pueden divulgar ni utilizar información, documentos o bio-especímenes que puedan identificarlo en cualquier ámbito civil, penal, administrativo, legislativo, federal, estatal o local. u otra acción, demanda o procedimiento, o ser utilizado como evidencia a menos que usted haya dado su consentimiento para este uso. La información, los documentos o las muestras biológicas protegidos por este Certificado no se pueden divulgar a ninguna otra persona que no esté relacionada con la investigación, a menos que exista una ley federal, estatal o local que exija la divulgación (por ejemplo, para denunciar abuso infantil, abuso de ancianos, intención de dañarse a sí mismo o a otros, o enfermedades transmisibles), usted ha dado su consentimiento para la divulgación, incluso para su tratamiento médico; o se utiliza para otras investigaciones científicas, según lo permitan las regulaciones federales que protegen a los sujetos de investigación.

El Certificado no se puede utilizar para rechazar una solicitud de información del personal de la agencia gubernamental federal o estatal que patrocina el proyecto y la cual es necesaria para la auditoría o evaluación del programa por parte del Instituto Nacional sobre el Abuso de Drogas (INAD) que está financiando el proyecto o para información que debe divulgarse para cumplir con los requisitos de la Administración de Alimentos y Medicamentos (FDA). También debe comprender que el Certificado de Confidencialidad no le impide divulgar voluntariamente información sobre usted o su participación en esta investigación. Si desea que la información de su investigación se divulgue a una aseguradora, proveedor de atención médica o cualquier otra persona que no esté relacionada con la investigación, usted debe dar su consentimiento para permitir que la investigación se divulgue.

Bajo la ley de California, debemos reportar información sobre incidentes conocidos o razonablemente sospechosos de abuso o negligencia infantil, de adulto dependiente o anciano, incluyendo abuso o negligencia física, sexual, emocional y financiera. Si algún investigador tiene o recibe dicha información, se le puede solicitar que la comunique a las autoridades correspondientes.

## ¿A quién puede llamar si tiene preguntas?

Se le ha explicado este estudio y se han respondido sus preguntas. Si tiene otras preguntas o problemas relacionados con la investigación, puede comunicarse con la Dra. Strathdee

Sitio del Estudio: San Diego Página 9 of 9

de manera confidencial al 858-822-1952 (llamar por cobrar) o con la Dr. Harvey-Vera al 858-967-7521.

Puede llamar a la Oficina del Programa de Protección de Investigaciones Humanas al 858-246-HRPP (858-246-4777) para informarse sobre sus derechos como sujeto de investigación o para informar problemas relacionados con la investigación.

| $\sim$ | ~ | | ,• • , |
|--------|---------|-----|----------------|
| 111 | tivno a | 111 | CONCONTIMIONTO |
| Ŋи | ummu | v | consentimiento |
| | , | ., | |

Ha recibido una copia de este documento de consentimiento.

| Usted Acepta participar. | |
|-------------------------------------------------------------------|-------|
| Firma del sujeto | Fecha |
| Firma de la persona que orienta sobre el consentimiento informado | Fecha |

# University of California, San Diego Consent to Act as a Research Subject

"LinkUP": A behavioral intervention within the project "Ethno-epidemiology of Hepatitis C (HCV), HIV and Overdose associated with Drug Markets and Drug Tourism", otherwise known as "La Frontera".

#### Introduction

Steffanie Strathdee, Ph.D. and the Harm Reduction Coalition of San Diego (HRCSD, "OnPoint") are conducting this research and asking for your consent to participate. This study is funded by the National Institutes of Health (NIH) and the Rapid Acceleration in Diagnostics in Underserved Populations (RADx-UP). This section provides a summary of important information. The rest of the form provides additional details.

- Research is voluntary- whether or not you join is your decision. You can discuss your decision with others (such as family and friends).
- You can say yes but change your mind later.
- If you say no, we will not hold your decision against you.
- Your decision will not affect any other benefits you may be entitled to.
- Please ask questions or mention concerns before, during or after the research.

**Summary:** We are conducting this research study to see if combining education, motivational interviewing (MI) and problem-solving increases uptake of COVID-19 testing and COVID-19 vaccination among people who inject drugs at syringe exchange programs. You will be asked to participate in a brief educational and/or behavioral session, and then offered free COVID-19 tests and referred to a nearby clinic who can offer COVID-19 vaccine. You will also be asked to complete one supplementary interview.

**Benefits:** Your participation in this study may help us to learn why some people delay COVID-19 testing or vaccination and about the effects of COVID-19 among people who inject drugs. We hope to use this information to conduct behavioral and health-related research among people who inject drugs, which may eventually be used to design appropriate and effective interventions and health programs in your community.

**Risks:** The most commonly expected risks of the study are discussing topics that might make you feel uncomfortable or upset. You can ask any of the researchers or OnPoint counselors to leave or stop talking to you at any time and change your mind about agreeing to participate in LinkUP even after we have started. If you would like to see a counselor after talking with us, we can arrange for that without any cost for you.

The most serious risks of the study may include loss of confidentiality. Although at no time will individual results or responses containing your name be available to persons

outside the study, there is a small chance that someone may discover that you participated in this study. If this were to happen, it could affect your employability and/or insurability. Our study team members will make every effort to protect your confidentiality and will make appropriate referrals to local health authorities for care. We will also provide you a study card and a 1-800 number so that our staff can advocate on your behalf if needed.

Study participants will be asked to provide their name, address and other personally identifying information to communicate and locate participants for follow-up visits or results from tests. This "locator" form is kept under locked cabinets at the study offices and only accessible to study staff. The information contained in the locator forms will not be shared with RADx\_UP or OnPoint staff.

Additional, detailed information about this research is provided below. Please feel free to ask questions before signing this consent.

#### What is the NIH and RADx-UP?

The NIH stands for the National Institutes of Health. The NIH is part of the United States Department of Health and Human Services. The NIH's purpose is to find new knowledge that will lead to better health for everyone. The NIH funded (provided support) for the RADx-UP program. We are calling the San Diego part of the study LinkUP.

RADx-UP is a health research program to learn more about COVID-19. If you join Link-UP, we will gather some data (information) about you. We will combine these with data from other people who join RADx-UP without your name or any identifying information attached that could identify you. We will study the data from all who join to understand how to help more people at risk for or with COVID-19.

# Why you have been asked to participate, how you were selected, and what is the approximate number of participants in the study?

You are being asked to participate in LinkUP because you are enrolled in the main La Frontera project, you are: a) at least 18 years old; b) you are resident of San Diego County where this study is taking place; c) you indicated in your follow up survey that you never voluntarily tested for COVID-19 outside of La Frontera; d) you have had two or fewer doses of COVID-19 vaccine, with your last dose being more than 6 months ago; e) you have agreed to share your medical records with the LinkUP study team; and f) have agreed to be contacted for this study. 149 other persons will be invited to participate in LinkUP.

# What will happen to you in this study and which procedures are standard of care and which are experimental?

If you decide to join the LinkUP study and if you completed your last study visit at La Frontera more than 3 months ago, La Frontera staff will ask you to participate in an interview that asks questions about your lifestyle, attitudes, behaviors, health issues and

whether or not you have had a COVID test or vaccine. You will be compensated \$20 for this visit.

Next, La Frontera staff will then give you a laminated coupon with the address and schedule for a nearby site of the OnPoint Syringe Exchange Program. Attending the OnPoint is voluntary. OnPoint is a syringe exchange program that offers free services at several locations around San Diego County, which includes free COVID-19 testing and referral to vaccination sites as part of standard of care. Four of these sites are participating in the LinkUP study. At two of the 4 sites, LinkUP participants will be offered COVID-19 education only, and at the other 2 sites, LinkUP participants will be offered COVID-19 and motivational interviewing (MI) counseling.

If you visit OnPoint, their staff will assign you a unique identifier (ID) if you have never used their program before. These IDs are generated using 1&3 letters of both first and last name, DOB, and a gender identifier M-1, F-2, Other-3.

OnPoint peer counselors will ask you a short 5 minute interview about COVID-19, including information about any symptoms (a change in your health) and test results. If you have a positive COVID-19 test, they will ask information about contact tracing (people who may have come in contact with you while you had COVID-19). They will ask about your medical history and if you have or have not had vaccines and why. Then, the OnPoint peer counselor will tell you about COVID-19, including information about the virus, how it is spread, what kinds of health problems it causes and what vaccines and treatments are available for it. They will tell you whether some information you may have heard about COVID-19 or COVID vaccines is correct and which is not. Depending on which OnPoint location you are visiting, the counselor may ask you to discuss any concerns about COVID-19 and vaccination with them. The OnPoint counselor will answer any questions you may have. No matter which OnPoint location you visit, this session will be completed within 45 minutes.

COVID-19 testing will be offered to you by the counselor as standard of care. You can refuse to participate in the LinkUP intervention and still have access to free rapid COVID-19 antigen tests (BiNaxNow® at syringe exchange programs across California, including OnPoint by the California Public Health Department (CPHD). You will be referred to a nearby clinic for free COVID-19 vaccination.

If you decide to get the rapid COVID-19 antigen test, the counselor will tell you your results in 15 minutes. If you test positive, you will be asked to provide a nasal swab for a PCR confirmatory test. You can refuse to have this test done if you don't want it. PCR testing of your nasal swab will be done at a certified lab within the next few days. If you give your contact information to the counselor, they will contact you to share the results of this test. If you test positive for COVID-19 on either of these tests or have symptoms, you will be referred to your medical provider for follow-up and you should isolate away from others. If you feel you have no safe place to isolate yourself, the counselor may

refer you to a shelter. If you test negative for the virus that causes COVID-19, the virus was not detected. However, it is possible to receive a false negative test result so you still might have COVID-19. If you are concerned you might have COVID-19 the counselor will refer you to a medical provider

If you decide to get an FDA-approved COVID-19 vaccine such as Pfizer, Moderna and Janssen you can get more information on where to get it from the OnPoint staff. The vaccine is given as a needle (shot) in your arm.

## How much time will each study procedure take?

If you completed your last La Frontera follow-up visit more than 3 months ago and now have to complete a behavioral survey, this process will take ~60 minutes. The OnPoint intake interview will take 10 minutes. The LinkUP counseling session will take ~45 minutes.

If you decide to get tested for COVID-19 as part of standard of care, the rapid test takes 15 minutes and you will get your test results on the spot. If you decide to get a COVID-19 PCR test, the nasal swabbing for the PCR test takes 3 minutes but you won't get your results for a few days. If you share your contact information with OnPoint staff, they will contact you so you can get your COVID-19 PCR test results.

# What will you do with my data?

We will gather data (information) about your counseling session, whether you got tested for COVID at the OnPoint syringe exchange site and whether you received a COVID-19 vaccination after your visit at OnPoint. We will gather some of these data from you directly which will be shared with La Frontera staff. To protect your confidentiality, a record linkage will be done without using name information (i.e., only based on your date of birth and gender, the combination of which is unique to you).

We may gather some of the data from other places where you may later receive a COVID-19 test, vaccine or treatment. Examples of the information that we may collect from you or other places include, but are not limited to the Harm Reduction Coalition of San Diego/OnPoint, San Diego Health and Human Services COVID-19 database, accessing your electronic health records from hospitals or drug treatment programs, and Centers for Medicare and Medicaid Services, among others.

Although your data will not be linked to your name, we will keep your data securely (which means with extra protection), along with the data from all the other people who take part in other RADx-UP programs around the country. Researchers will use the data to learn more about COVID-19 or other diseases and conditions.

The Duke Clinical Research Institute (DCRI) is a research group chosen by the National Institute of Health (NIH) to combine the data collected from everyone taking part in RADx-UP studies.

Page **5** of **8** 

The DCRI will build a RADx-UP database (system that hold electronic information) that will hold all the non-identifiable information you agree to give.

- You will be assigned a study code and you will only be identified in this database by this study code.
- It will not contain your name or other information that could easily identify you.
- We plan to transfer and keep these non-identifiable data in a secure database for COVID19 research at the NIH. Other researchers may use these data for studies, other than the ones stated in this consent form.
- Researchers will only have access to your non-identifiable data and cannot link the data back to you.
- Because the data cannot be linked back to you, we will not contact you to inform you or ask your permission before sharing the data with researchers.

I agree to let OnPoint and La Frontera link my identifiable and non-identifiable data without using my name.

| Yes | No |
|----------|-----------------|
| Initials | <u>Initials</u> |

#### What risks are associated with this study?

There is the potential for the loss of confidentiality. Although at no time will individual results or responses to questions be available to persons outside the study and study forms will not contain your name, there is a small chance that someone may discover that you participated in this study. The personally identifying information such as name and address contained in the locator forms will be kept under locked separate cabinets at the study offices at all times only available to study staff. It is also your choice whether or not to tell people that you have taken part in this study. There is also a very small chance that someone could learn the answers you have given to the questions asked in the LinkUP intervention. If this were to happen, it could affect your employability and/or insurability.

Because this is a research study, there may also be some unknown risks that are currently unforeseeable. You will be informed of any significant new findings.

## What are the alternatives to participating in this study?

Alternatives to this study are to not participate. It is your decision to join the study or not. You can drop out of this study at any time. If you ever don't want to answer a specific question you do not have to. If you withdraw from the study you will be asked by Dr. Harvey-Vera or Dr. Strathdee whether you wish to take back your consent to use

information gathered up to that point. You may inspect and make a copy of the records of your participation in this project. You can refuse to participate in the LinkUP intervention and still have access to free rapid COVID-19 antigen tests (BiNaxNow®) and to syringe exchange programs across California, including OnPoint by the California Department of Public Health (CDPH).

## What happens if you change your mind about participating?

You can withdraw from the study at any time. If you decide that you no longer wish to continue in this study, you will be asked by Dr. Harvey-Vera or Dr. Strathdee whether you wish to take back your consent to use information gathered up to that point. You may inspect and make a copy of the records of your participation in this subject. You will be told if any important new information is found during the course of this study that may affect your wanting to continue.

## Can you be withdrawn from the study without your consent?

Due to the nature of scientific research, the researcher may withdraw you from the study at any time. You may also be withdrawn from the study if you do not follow the instructions given you by the study personnel.

## Will you be compensated for participating in this study?

If you need to complete the behavioral survey, you will be compensated \$20 upon completion of your LinkUP interview. You will be compensated \$10 for your visit to OnPoint.

## Are there any costs associated with participating in this study?

There will be no cost to you for participating in this study.

## What if you are injured as a direct result of being in this study?

If you are injured as a direct result of participation in this research, the University of California will provide any medical care you need to treat those injuries. The University will not provide any other form of compensation to you if you are injured. You may call the Human Research Protections Program Office at 858-246-HRPP (858-246-4777) for more information about this, to inquire about your rights as a research subject or to report research-related problems.

### How will you protect my privacy?

Your privacy is very important to us. We will take great care to protect your privacy. However, there is always a chance that, even with our best efforts, your identity and/or information collected during this study may be accidentally released or seen by unauthorized persons. Here are a few steps we will take:

• Everyone working on this study has been trained to respect the privacy of study participants. They will never discuss what you have told them in a way that could identify you.

- Your name or other identifying information contained in the locator forms will not be on any notes or data. This consent form and the locator form will be the only form with your name on it. It will be stored at the University of California, San Diego, in La Jolla CA in a locked drawer. We will never reveal that you participated or any other information about your visit to anyone else as far as the law will allow us. Your survey information will be labeled only with a study number and not your name.
- Data will be stored on protected, secure and encrypted computer systems. We will limit and keep track of who can see these data. Our study team will use computers managed by our UCSD Health IT department, equipped with malware and antivirus software, TPM security chips, and will operate on a VPN.
- Anyone who can see these data will have to use a password.
- We will take steps to protect your information from others that should not be able to see it.
- When your data are shared with other researchers, they will not have information that can identify you.
- After such removal, the information could be used for future research studies or distributed to another investigator for future research studies without your additional informed consent.

This research will be covered by a Certificate of Confidentiality from the United States Government. Researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research *unless* there is a federal, state, or local law that requires disclosure (such as to report child abuse, elder abuse, intent to hurt self or others, or communicable diseases), you have consented to the disclosure, including for your medical treatment; or it is used for other scientific research, as allowed by federal regulations protecting research subjects.

The Certificate cannot be used to refuse a request for information from personnel of federal or state government agency sponsoring the project that is needed for auditing or program evaluation by the National Institute on Drug Abuse (NIDA) which is funding the project or for information that must be disclosed in order to meet the requirements of the Food and Drug Administration (FDA). You should also understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the research to release it.

Under California law, we must report information about known or reasonably suspected incidents of abuse or neglect of a child, dependent adult or elder including physical, sexual, emotional, and financial abuse or neglect. If any investigator has or is given such information, he or she may be required to report such information to the appropriate authorities.

## Who can you call if you have questions?

Your Signature and Consent

This study has been explained to you and your questions have been answered. If you have other questions or research-related problems, you may reach Dr. Strathdee confidentially at 858-822-1952 (call collect) or Dr. Harvey-Vera at 858-967-7521.

You may call the Human Research Protections Program Office at 858-246-HRPP (858-246-4777) to inquire about your rights as a research subject or to report research-related problems.

| You have received a copy of this consent document. | |
|---|---|
| You agree to participate. | |
| Subject's signature | Date |
| Signature of the person conducting the informed consent discussion | Date |